CLINICAL TRIAL: NCT04516434
Title: AMPLIFY: Amplifying Sensation in Underactive Bladder
Brief Title: Amplifying Sensation in Underactive Bladder
Acronym: AMPLIFY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00106457
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Urinary Bladder, Underactive
Keywords: electrical stimulation; urodynamics; bladder; urethra
MeSH Terms: conditions — Urinary Bladder, Underactive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Intraurethral Electrical Stimulation (Experimental): This procedure is specific to the urethral stimulation arm. A sterile stimulation catheter (custom, 7-French) will be placed in the urethra and positioned with the electrode contact 10-14 mm from the bladder neck to stimulate the proximal urethra. A single return electrode will also be placed on the abdominal skin above the pubic bone. Stimuli will be delivered as 0.2 ms charge-balanced biphasic rectangular current pulses. Stimulation frequency will be 2-20 Hz and amplitude will be adjusted individually to 80% of the maximum tolerable intensity. Electrical stimulation will be applied to the proximal urethra at "strong desire to void" during cystometry. The participant will then be given permission to void at "maximum cystometric capacity" with continuous intraurethral stimulation.
  Interventions: Device: Neurometer Neurotron CPT; Procedure: Cystometry; Procedure: Pressure-flow study
- Intravesical Electrical Stimulation (Experimental): This procedure is specific to the bladder stimulation arm. A sterile stimulation catheter (custom, 7-French) will be placed in the bladder through the urethra and the electrode contacts will be positioned to be floating within the bladder. A single return electrode will also be placed on the abdominal skin above the pubic bone. Stimuli will be delivered as 0.2 ms charge-balanced biphasic rectangular current pulses. Stimulation frequency will be set at 20 Hz and amplitude will be adjusted individually to 80% of the maximum tolerable intensity. Electrical stimulation will be applied to bladder sensory nerves for up to 60 minutes prior to the start of urodynamic studies.
  Interventions: Device: Neurometer Neurotron CPT; Procedure: Cystometry; Procedure: Pressure-flow study

INTERVENTIONS:
Device: Neurometer Neurotron CPT — All participants will undergo CPT testing. A Neurotron catheter (12-French) with electrode will be inserted through the urethra into the bladder. The catheter balloon will be inflated and positioned at the urethrovesical junction to stimulate the urethra 10-14 mm from the bladder neck. For bladder stimulation, the catheter balloon will be deflated and the catheter will be advanced into the bladder. The device will deliver sine wave stimulus pulses at 5, 250, and 2,000 Hz. CPT will be established using an automated forced choice paradigm by the method of levels. Testing order of the bladder and urethra will be randomized between participants.
Procedure: Cystometry — After bladder stimulation or during intraurethral stimulation, cystometry will be performed to assess bladder sensation and storage. A dual-chamber 8-French catheter will be passed through the urethra into the bladder for retrograde filling. A second 8-French catheter will be placed in the vagina to measure intra-abdominal pressure. A stimulation electrode catheter will only be inserted in the intraurethral stimulation arm. EMG pads will then be placed at 3 and 9 o'clock on each side of the perineum. The bladder will then be filled with room-temperature sterile saline solution in a retrograde fashion using a pump. Bladder sensation and urgency will be assessed while filling.
Procedure: Pressure-flow study — A pressure flow study will be performed to evaluate voiding function after stimulation. The transurethral and intra-vaginal catheters are left in place after cystometry and the participant will be asked to void around them, into a commode. Bladder and abdominal pressures will be recorded, as well as urine flow over time.

SUMMARY:
The purpose of this study is to determine the influence of intravesical (bladder) electrical stimulation and intraurethral electrical stimulation on bothersome symptoms and bladder function in neurologically-intact adult women with underactive bladder. The investigators hypothesize that electrical stimulation will decrease bothersome urinary symptoms relative to baseline and increase voided percentage during pressure-flow studies compared to their routine clinical exam.

DETAILED DESCRIPTION:
1. Objective: The overall objective of this study is to improve lower urinary tract symptoms (LUTS) in adult neurologically-intact women with underactive bladder through electrical stimulation of bladder sensory nerves or urethral sensory nerves.
2. Background and Significance: The storage and elimination of urine is regulated by neural circuits in the brain and spinal cord to coordinate function between the urinary bladder and the urethra. During micturition (bladder emptying), the elimination of urine is facilitated by bladder muscle (detrusor) contraction and urethral and pelvic floor muscle relaxation. Urine flow through the urethra also activates sensory nerves to amplify bladder contractions and maintain efficient bladder emptying. Incomplete emptying and urinary retention occur when these mechanisms are disrupted or poorly coordinated.

   Incomplete emptying due to underactive bladder is a poorly understood health concern that symptomatically affects up to 40% of the population, with the highest prevalence of symptoms in older men and women. Despite the high prevalence of symptoms, the diagnosis of an underactive bladder remains low due to the lack of consistent terminology and standardized diagnostic criteria. This results in defining underactive bladder by a symptom complex that may involve reduced motor drive (detrusor underactivity) during bladder emptying and/or reduced sensory drive during filling and emptying. Symptoms experienced by persons with underactive bladder include nocturia, urinary frequency, urgency, incontinence, slow stream, hesitancy, straining, and sensation of incomplete emptying. The most common symptoms are nocturia, slow stream, frequency, hesitancy, and the impact of these symptoms on quality of life is substantial for many patients.

   The management options for persons with underactive bladder include double-void, intermittent self-catheterization, or pharmacotherapy. However, these treatments are associated with poor quality of life and patients often fail to completely resolve the lower urinary tract symptoms (LUTS). There is a need to clarify the pathological mechanisms underlying underactive bladder to improve therapeutic outcomes. One approach to clarify reduced sensory drive is to evaluate the functional integrity of sensory nerves with quantitative sensory testing. Current perception threshold (CPT) testing delivers electrical stimulation to activate nerve fibers that evoke sensory perception, and changes in bladder sensory pathways were demonstrated in persons with diabetic detrusor underactivity. These diagnostic tests, however, have not been applied to neurologically intact adult women with underactive bladder and may provide insight into pathological sensory dysfunction.

   The proposed research will quantify sensory nerve sensitivity in the bladder and urethra in adult women with underactive bladder. The investigators will then amplify sensory nerve activity via continuous electrical stimulation to improve LUTS associated with underactive bladder. Achieving the proposed objectives will establish a prognostic marker for rationally guided electrical stimulation in women with underactive bladder. Understanding how these mechanisms contribute to impaired emptying in underactive bladder will enable the development of novel therapeutics to enhance quality of life.
3. Subject Recruitment: Established patients with underactive bladder will be identified by MaestroCare chart review. New patients with underactive bladder will be identified by Duke urogynecologists who see patients at one of two urogynecologic offices (Navaho Clinic in Raleigh or Patterson Place in Durham).
4. Design and Procedures: The investigators will perform a parallel interventional study with two non-randomized study arms (bladder stimulation and urethral stimulation). Potential participants will be screened remotely by email via RedCap by completing a questionnaire to determine bothersome symptoms and perceptions of bladder function. Potential participants that meet eligibility criteria will be scheduled for an in person study procedure visit, where informed consent will be signed. Participants will then undergo current perception threshold (CPT) testing, where electrical stimulation will be delivered via a catheter to the urethra (intraurethral) and bladder (intravesical) to evoke sensation. The CPT results will inform whether the participant receives an investigational session of intravesical (bladder) electrical stimulation or intraurethral electrical stimulation. Following electrical stimulation, the participant will undergo urodynamic studies (cystometrogram, pressure-flow study) to assess bladder function after the investigational stimulation procedures. The participant will also be asked to complete remotely by email a post-study symptom RedCap questionnaire 7 days after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18 and older
* Able to provide informed consent and agree to the study risks
* Willing to withdraw from medications affecting urination for the 48 hours prior to the procedure (e.g., alpha-adrenergic antagonists, cholinergic agonists, cholinesterase inhibitors)
* Has the below response to 2 of the 3 questions:

  1. Questions regarding self-reported poor sensation during bladder filling or emptying (one or more of the below)

     * In the past 7 days, where did the participant feel sensations when needing to urinate? Answer: "No" response for Bladder Area
     * In the past 7 days, how often did the participant have no sensation of urine flow while urinating? Answer: "Most of the time" or "Every time" response
     * In the past 7 days, how often did the participant feel that the bladder was not completely empty after urination? Answer: "Most of the time" or "Every time" response
  2. Questions regarding self-reported bothersome urinary symptoms (one or more of the below)

     * In the past 7 days, how satisfied was the participant with bladder function? Answer: "Not at all satisfied" or "Somewhat satisfied" response
     * In the past 7 days, how bothered was the participant by urinary symptoms? Answer: "Very bothered" or "Extremely bothered" response
  3. Standard uroflowmetry with a voiding efficiency (voided volume / voided volume + residual volume) of < 80%, voided volume + residual volume must be >150ml for measurement

Exclusion Criteria:

* Preexisting neurological impairment (e.g., spinal cord injury, multiple sclerosis, Guillain-Barre, cauda equina syndrome, cerebrovascular accident, Parkinson's disease, traumatic brain injury)
* Functional obstruction demonstrated by either elevated pelvic floor activity on EMG during standard pressure flow study or high tone pelvic floor on clinical exam)
* Pelvic organ prolapse beyond introitus
* Active urinary tract infection (candidate would be deferred until treated)
* Positive pregnancy test
* Less than 6 weeks postpartum
* Unevaluated hematuria
* Urethral stricture/stenosis
* Surgical obstruction i.e., urinary retention due to obstructive sling or other anti incontinence procedure
* Surgical procedures to increase bladder capacity (e.g., augmentation cystoplasty)
* Active sacral neuromodulation or ongoing posterior tibial nerve stimulation sessions
* Botulinum toxin injection in the past six months
* History of genitourinary or gastrointestinal cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Amundsen, MD, Study Chair — Duke University; Em Abbott, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Plaza Patterson Place, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowler CJ, Griffiths D, de Groat WC. The neural control of micturition. Nat Rev Neurosci. 2008 Jun;9(6):453-66. doi: 10.1038/nrn2401. PMID 18490916
- [Background] Jung SY, Fraser MO, Ozawa H, Yokoyama O, Yoshiyama M, De Groat WC, Chancellor MB. Urethral afferent nerve activity affects the micturition reflex; implication for the relationship between stress incontinence and detrusor instability. J Urol. 1999 Jul;162(1):204-12. doi: 10.1097/00005392-199907000-00069. PMID 10379788
- [Background] Bump RC. The urethrodetrusor facilitative reflex in women: results of urethral perfusion studies. Am J Obstet Gynecol. 2000 Apr;182(4):794-802; discussion 802-4. doi: 10.1016/s0002-9378(00)70328-0. PMID 10764455
- [Background] Osman NI, Chapple CR, Abrams P, Dmochowski R, Haab F, Nitti V, Koelbl H, van Kerrebroeck P, Wein AJ. Detrusor underactivity and the underactive bladder: a new clinical entity? A review of current terminology, definitions, epidemiology, aetiology, and diagnosis. Eur Urol. 2014 Feb;65(2):389-98. doi: 10.1016/j.eururo.2013.10.015. Epub 2013 Oct 26. PMID 24184024
- [Background] Jeong SJ, Kim HJ, Lee YJ, Lee JK, Lee BK, Choo YM, Oh JJ, Lee SC, Jeong CW, Yoon CY, Hong SK, Byun SS, Lee SE. Prevalence and Clinical Features of Detrusor Underactivity among Elderly with Lower Urinary Tract Symptoms: A Comparison between Men and Women. Korean J Urol. 2012 May;53(5):342-8. doi: 10.4111/kju.2012.53.5.342. Epub 2012 May 18. PMID 22670194
- [Background] Chapple CR, Osman NI, Birder L, van Koeveringe GA, Oelke M, Nitti VW, Drake MJ, Yamaguchi O, Abrams P, Smith PP. The underactive bladder: a new clinical concept? Eur Urol. 2015 Sep;68(3):351-3. doi: 10.1016/j.eururo.2015.02.030. Epub 2015 Mar 11. PMID 25770481
- [Background] Gammie A, Kaper M, Dorrepaal C, Kos T, Abrams P. Signs and Symptoms of Detrusor Underactivity: An Analysis of Clinical Presentation and Urodynamic Tests From a Large Group of Patients Undergoing Pressure Flow Studies. Eur Urol. 2016 Feb;69(2):361-9. doi: 10.1016/j.eururo.2015.08.014. Epub 2015 Aug 28. PMID 26318706
- [Background] Uren AD, Cotterill N, Harding C, Hillary C, Chapple C, Klaver M, Bongaerts D, Hakimi Z, Abrams P. Qualitative Exploration of the Patient Experience of Underactive Bladder. Eur Urol. 2017 Sep;72(3):402-407. doi: 10.1016/j.eururo.2017.03.045. Epub 2017 Apr 8. PMID 28400168
- [Background] Miyazato M, Yoshimura N, Chancellor MB. The other bladder syndrome: underactive bladder. Rev Urol. 2013;15(1):11-22. PMID 23671401
- [Background] Ukimura O, Ushijima S, Honjo H, Iwata T, Suzuki K, Hirahara N, Okihara K, Mizutani Y, Kawauchi A, Miki T. Neuroselective current perception threshold evaluation of bladder mucosal sensory function. Eur Urol. 2004 Jan;45(1):70-6. doi: 10.1016/j.eururo.2003.08.004. PMID 14667519
- [Background] Kenton K, Simmons J, FitzGerald MP, Lowenstein L, Brubaker L. Urethral and bladder current perception thresholds: normative data in women. J Urol. 2007 Jul;178(1):189-92; discussion 192. doi: 10.1016/j.juro.2007.03.032. Epub 2007 May 17. PMID 17499783
- [Background] Lee WC, Wu HP, Tai TY, Yu HJ, Chiang PH. Investigation of urodynamic characteristics and bladder sensory function in the early stages of diabetic bladder dysfunction in women with type 2 diabetes. J Urol. 2009 Jan;181(1):198-203. doi: 10.1016/j.juro.2008.09.021. Epub 2008 Nov 14. PMID 19013605
- [Background] Cella D, Smith AR, Griffith JW, Flynn KE, Bradley CS, Gillespie BW, Kirkali Z, Talaty P, Jelovsek JE, Helfand BT, Weinfurt KP; LURN Study Group. A new outcome measure for LUTS: Symptoms of Lower Urinary Tract Dysfunction Research Network Symptom Index-29 (LURN SI-29) questionnaire. Neurourol Urodyn. 2019 Aug;38(6):1751-1759. doi: 10.1002/nau.24067. Epub 2019 Jun 21. PMID 31225927
- [Background] Gladh G, Mattsson S, Lindstrom S. Intravesical electrical stimulation in the treatment of micturition dysfunction in children. Neurourol Urodyn. 2003;22(3):233-42. doi: 10.1002/nau.10078. PMID 12707874
- [Background] Jiang CH, Lindstrom S. Optimal conditions for the long-term modulation of the micturition reflex by intravesical electrical stimulation: an experimental study in the rat. BJU Int. 1999 Mar;83(4):483-7. doi: 10.1046/j.1464-410x.1999.00947.x. PMID 10210575
- [Background] Deng H, Liao L, Wu J, Chen G, Li X, Wang Z, Wan L. Clinical efficacy of intravesical electrical stimulation on detrusor underactivity: 8 Years of experience from a single center. Medicine (Baltimore). 2017 Sep;96(38):e8020. doi: 10.1097/MD.0000000000008020. PMID 28930838
- [Background] Gustafson KJ, Creasey GH, Grill WM. A urethral afferent mediated excitatory bladder reflex exists in humans. Neurosci Lett. 2004 Apr 22;360(1-2):9-12. doi: 10.1016/j.neulet.2004.01.001. PMID 15082166
- [Background] Yoo PB, Horvath EE, Amundsen CL, Webster GD, Grill WM. Multiple pudendal sensory pathways reflexly modulate bladder and urethral activity in patients with spinal cord injury. J Urol. 2011 Feb;185(2):737-43. doi: 10.1016/j.juro.2010.09.079. Epub 2010 Dec 18. PMID 21168860

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravesical Electrical Stimulation: To evaluate improvement of sensations during bladder filling and emptying with electrical stimulation to the bladder or urethra. The researchers will use the values obtained from investigational sensory testing to deliver continuous electrical stimulation to the bladder . The location depends on which value is higher compared to normal. A nurse or doctor will place a catheter with electrodes to perform this investigational study procedure to the bladder (up to 60 minutes). The researchers will also place a surface patch on the participant's abdomen to disperse the electrical current and reduce discomfort.
- Intraurethral Electrical Stimulation: To evaluate improvement of sensations during bladder filling and emptying with electrical stimulation to the bladder or urethra. The researchers will use the values obtained from investigational sensory testing to deliver continuous electrical stimulation to the urethra. The location depends on which value is higher compared to normal. A nurse or doctor will place a catheter with electrodes to perform this investigational study procedure to the urethra (up to 15 minutes). Two surface patches (electrodes) will be placed at the 3 o'clock and 9 o'clock positions, 1 to 3 centimeters from the around the vaginal opening. These electronic sensors will record muscle activity while the bladder is contracting.
  The intraurethral stimulation will occur during routine urodynamic evaluation when the participant urinates on a special toilet.
Period: Overall Study
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6) | 67 (4) | 68 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Voiding Efficiency
Description: Use of intraurethral electrical stimulation or intravesical electrical stimulation to assess increase in voided percentage during pressure-flow studies. Voiding efficiency is calculated as voided volume divided by the sum of voided volume and residual volume.
Time Frame: Baseline, pressure-flow study (up to 60 minutes)
Measure: Mean (Standard Deviation); unit: voided percentage
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
Number analyzed (Participants) | 12 | 8
voided percentage
  Baseline | 32 (31) | 53 (22)
  Pressure-flow study (up to 60 minutes) | 43 (37) | 46 (27)
Statistical Analysis 1: Comparison: Intravesical Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 1, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intraurethral Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 0.99, Mixed Models Analysis

2. Primary Outcome: Change in Bothersome Symptoms and Sensation
Description: Lower Urinary Tract Dysfunction Research Network Symptom Index-29 (LURN SI-29) to assess whether electrical stimulation decreases urinary bothersome symptoms and increases bladder sensation during filling and emptying. Scores range from 0 (least severe) to 100 (most severe). Higher scores indicate greater severity of lower urinary tract symptoms.
Time Frame: baseline and post study procedures, up to 60 minutes
Measure: Mean (Standard Deviation); unit: CASUS questionnaire scores
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
Number analyzed (Participants) | 12 | 8
CASUS questionnaire scores
  Baseline | 52 (15) | 53 (11)
  Post Study Procedures | 46 (16) | 39 (18)
Statistical Analysis 1: Comparison: Intravesical Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 0.08, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intraurethral Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 0.045, Mixed Models Analysis

3. Secondary Outcome: Current Perception Threshold
Description: Assess bladder or urethral current perception threshold (CPT) in women with underactive bladder compared to normative values. The CPT value determined by the device is defined as the average of the minimum amplitude of the stimulus consistently detected and the stimulus 40 µA lower that was consistently not detected.
Time Frame: CPT, up to 60 minutes
Measure: Mean (Standard Deviation); unit: mA (maximum amplitude)
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
Number analyzed (Participants) | 12 | 8
mA (maximum amplitude)
  5 Hz | 8.57 (3.23) | 8.27 (3.61)
  250 Hz | 9.99 (0.00) | 9.04 (0.40)
  2000 Hz | 9.99 (0.00) | 9.99 (0.00)

4. Secondary Outcome: Cystometry Volume
Description: Use of intravesical electrical stimulation to assess volumes during cystometry. Bladder sensation and urgency assessed at volume of first sensation during bladder filling, first desire to void, strong desire to void, and maximum cystometric capacity.
Time Frame: cystometry before stimulation and after stimulation (up to 60 minutes)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
Number analyzed (Participants) | 12 | 8
mL
  first sensation of bladder filling - before stimulation | 290 (159) | 253 (122)
  first sensation of bladder filling - after stimulation | 281 (146) | 357 (135)
  maximum cystometric capacity - before stimulation | 517 (263) | 458 (225)
  maximum cystometric capacity - after stimulation | 528 (253) | 646 (211)
Statistical Analysis 1: Comparison: Intravesical Electrical Stimulation; First sensation of bladder filling - change in cystometry before stimulation and after stimulation (up to 60 minutes); Test type: Other — Descriptive analysis; p = 1, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intraurethral Electrical Stimulation; First sensation of bladder filling - change in cystometry before stimulation and after stimulation (up to 60 minutes); Test type: Other — Descriptive analysis; p = 0.41, Mixed Models Analysis
Statistical Analysis 3: Comparison: Intravesical Electrical Stimulation; Maximum cystometric capacity - change in cystometry before stimulation and after stimulation (up to 60 minutes); Test type: Other — Descriptive analysis; p = 1, Mixed Models Analysis
Statistical Analysis 4: Comparison: Intraurethral Electrical Stimulation; Maximum cystometric capacity - change in cystometry before stimulation and after stimulation (up to 60 minutes); Test type: Other — Descriptive analysis; p = 0.01, Mixed Models Analysis

5. Secondary Outcome: Bladder Contraction Strength
Description: Use of intraurethral electrical stimulation to assess contraction strength relative to baseline. Bladder pressure (cmH2O) is recorded over time during voiding.
Time Frame: Baseline, pressure-flow study (up to 60 minutes)
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
Number analyzed (Participants) | 12 | 8
cmH2O
  Baseline | 11 (32) | 33 (41)
  Pressure-flow study (up to 60 minutes) | 21 (18) | 25 (27)
Statistical Analysis 1: Comparison: Intravesical Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 1, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intraurethral Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 1, Mixed Models Analysis

6. Secondary Outcome: Bladder Contraction Duration
Description: Use of intraurethral electrical stimulation to assess flow duration during a bladder contraction relative to baseline.
Time Frame: Baseline, pressure-flow study (up to 60 minutes)
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
Number analyzed (Participants) | 12 | 8
mL/s
  Baseline | 8 (3) | 15 (3)
  Pressure-flow study (up to 60 minutes) | 15 (12) | 13 (7)
Statistical Analysis 1: Comparison: Intravesical Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 1, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intraurethral Electrical Stimulation; Change from baseline to after the pressure-flow study; Test type: Other — Descriptive analysis; p = 0.99, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: One month post study completion
Arm/Group | Intravesical Electrical Stimulation | Intraurethral Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 3/12 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravesical Electrical Stimulation (N=12) | Intraurethral Electrical Stimulation (N=8)
Urinary tract infection (Renal and urinary disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04516434/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04516434/ICF_000.pdf